CLINICAL TRIAL: NCT01646619
Title: A Multicenter Randomized Controlled Trial of Therapeutic Hypothermia Plus Magnesium Sulphate (MgSO4) Versus Therapeutic Hypothermia Plus Placebo in the Management of Term and Near Term Babies With Hypoxic Ischemic Encephalopathy
Brief Title: Efficacy Study of Hypothermia Plus Magnesium Sulphate(MgSO4) in the Management of Term and Near Term Babies With Hypoxic Ischemic Encephalopathy
Acronym: MagCool
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sajjad Rahman (Industry)
Responsible Party: Sponsor-Investigator, Sajjad Rahman, Senior Consultant Perinatal Medicine, Hamad Medical Corporation
Organization: Hamad Medical Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GC 1028A; HMC-GC1028A (Other: Hamad Medical Corporation)
Record Dates: First submitted 2012-07-05; First posted 2012-07-20 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Severe Hypoxic Ischemic Encephalopathy; Moderate Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic Ischemic Encephalopathy; Therapeutic Hypothermia; Therapeutic Hypothermia plus Adjuvant Therapy; Cooling
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Magnesium Sulfate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia + Magnesium Sulphate (Active Comparator)
  Interventions: Drug: Magnesium Sulphate
- Hypothermia+ Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Sulphate — 10% MgSo4 (100mg/ml) given in a dose of 250mg/kg IV q 24 hrly for 3 doses(2.5ml/kg).
  Diluent: Dextrose 5%.
  Other Names: MgSo4
  Arms: Hypothermia + Magnesium Sulphate
Drug: Placebo — Normal Saline 0.9% Sodium Chloride is diluted in 5% Dextrose to be given as 2.5ml/kg IV q24 hrly for 3 doses.
  Other Names: Normal Saline; 0.9% Sodium Chloride
  Arms: Hypothermia+ Placebo

SUMMARY:
The purpose of this study is to assess whether the addition of a drug such as Magnesium sulphate while providing therapeutic hypothermia (or cooling) to babies who are asphyxiated at birth provides additional benefit to the babies' survival and outcome compared to cooling alone.

DETAILED DESCRIPTION:
Perinatal Asphyxia continues to be a major cause of neonatal mortality and morbidity even in the most technologically advanced and prosperous countries of the world. The incidence remains unchanged; 1-2% of live births in developed world countries and much higher in developing world countries. Perinatal Asphyxia is a multisystem disorder. Neonatal brain is the most important organ affected by Asphyxic insult because the resulting neuronal damage is permanent. Hypoxic Ischemic Encephalopathy (HIE), the pathognomonic clinical syndrome of asphyxic neuronal insult, occurs in 50-60% of babies with Perinatal Asphyxia. Moderate and severe HIE causes significant neonatal mortality and morbidity. Among patients with moderate HIE, 10-20% die and 30-40% develop neurological deficit, whereas 50% of patients with severe HIE die and almost all survivors develop neurological deficits. Hence the toll on the society continues to be very high in spite of dramatic improvements in neonatal intact survival, particularly in developed world countries.

Until recent years, the management of HIE was limited to supportive intensive care only because there was no specific treatment available to rescue neurons during HIE. However, over the last decade, therapeutic Hypothermia, has emerged as a promising new therapy in reducing neonatal mortality and morbidity due to HIE. This is due to improved understanding of the physiology of neuronal damage during asphyxia insult. Hypoxic Ischemic Encephalopathy (HIE) is a dynamic process which evolves over a period of seventy two hours starting from the time of insult. Two distinct episodes of neuronal damage occur during this time:

1. The immediate (primary) hypoxic insult followed by a
2. latent period of recovery which lasts for almost six hours.

This is followed by a much longer and profound period of secondary neuronal damage due to the release of chemical mediators. Therapeutic modalities which can potentially reduce the release of these chemical mediators will provide neuronal rescue. Moderate controlled hypothermia (33.5-34.5 0C) offered during the first 72 hours after the asphyxic insult is one such therapeutic modality which has been the subject of animal studies as well as extensive multicenter trails in human infants over the last two decades.

The studies on animal models have not only confirmed the safety of moderate therapeutic hypothermia; they have also shown a dramatic neuronal rescue in experimental HIE model of lambs subjected to prolonged therapeutic hypothermia immediately after birth. This was followed by pilot RCT's in human infants; the outcomes of which were very encouraging. However a universal change of practice requires large well designed multicenter trails and Meta analyses.

After having established therapeutic hypothermia as a safe and effective modality for neuroprotection in HIE, the neonatologists are facing a new question. Can the investigators enhance the neuroprotective effect of therapeutic hypothermia by adding other potential neuroprotective agents? These potential therapeutic agents include Xenon, Erythropoetin, Magnisium sulphate, Allopurinol, opoids, Topiramate, Inhaled Nitric Oxide (iNO), N-Acetylcystine, Minocycline and Melatonin.13,17 Due to their different mechanisms of action, it is likely that these neuroprotective therapies may add incrementally to the proven beneficial effects of hypothermia. Indeed hypothermia may buy additional time for these neuroprotective agents to act within an expanded 'therapeutic window'.13 These Hypothermia plus therapies are going to be the subject of many new RCT's worldwide over the next few years.

Magnesium Sulphate, a potential neuroprotective agent, acts by reducing neuronal excitotoxicity. MgSO4 has long been used in Obstertrics as a tocolytic agent and has a proven neuroprotective effect in preterm babies born to mothers tocolyzed with MgSO4. A recently conducted RCT in human neonates has compared postnatal magnesium sulfate with placebo in the management of Neonatal HIE. This study, which did not use hypothermia therapy due to lack of facilities, has shown that treatment with MgSO4 improves neurologic outcomes at discharge in term neonates with severe perinatal asphyxia. The animal studies done by Knuckley's group has compared a combination of therapeutic hypothermia and MgSO4 with therapeutic hypothermia alone. In their rat model MgSO4 alone had a minimal beneficial effect. However, MgSO4 plus hypothermia had a significant beneficial effect in reducing the size of the post asphyxia infarct. This animal focal stroke model provides an intriguing suggestion that hypothermia plus MgSO4 provides an additive neuroprotection. No human studies have been done so far to test the difference between therapeutic hypothermia alone and therapeutic hypothermia plus MgSO4. Mag Cool Study (Hypothermia plus MgSO4 Vs Hypothermia plus placebo) will test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

The babies will be assessed sequentially by criteria A, B and C listed below:

A. Evidence of Perinatal Asphyxia at birth: Infants ≥35 completed weeks gestation admitted to the NICU with at least one of the following:

1. Apgar score of <5 at 10 minutes after birth
2. Continued need for resuscitation, including endotracheal or mask ventilation, at 10 minutes after birth
3. Acidosis within 60 minutes of birth (defined as any occurrence of umbilical cord arterial or venous pH <7.00 or otherwise arterial or capillary pH <7.00)
4. Base Deficit (-16 mmol/L or more) in umbilical cord or any blood sample (arterial, venous or capillary) within 60 minutes of birth

Infants that meet criteria A will be assessed for whether they meet the neurological abnormality entry criteria (B) by trained personnel:

B. Clinical Evidence of Moderate to severe encephalopathy, consisting of altered state of consciousness (lethargy, stupor or coma) AND at least one of the following:

1. hypotonia
2. abnormal reflexes including oculomotor or pupillary abnormalities
3. absent or weak suck
4. clinical seizures

Infants who meet criteria A & B will be assessed by aEEG only in units where facility for Cerebral Function Monitoring (CFM) is available.

C. (Optional) At least 30 minutes duration of amplitude integrated EEG recording that shows abnormal background aEEG activity or seizures. There must be one of the following:

1. normal background with some seizure activity
2. continuous seizure activity
3. moderately abnormal activity: Only Lower border below 5 mV. upper border remains above 10mV
4. Severely Abnormal activity (suppressed activity): Both Lower border below 5 mV and upper border below 10mV

Exclusion Criteria:

* Infants expected to be > 6 hours of age at the time of randomization.Every effort will be made to ensure entry to the study before 3 hours of age.
* Major congenital abnormalities, such as diaphragmatic hernia requiring ventilation, or congenital abnormalities suggestive of chromosomal anomaly or other syndromes that includes brain dysgenesis.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Combined outcome of Mortality and Severe Neurodevelopmental Disability | 18 - 24 months of age
  Severe Neurodevelopmental Disability will be assessed at discharge from hospital and at 18-24 months of age to assess developmental delay and cerebral palsy using the Bayley Scale of Infant Development II.

SECONDARY OUTCOMES:
Persistent Hypotension | Duration of hypothermia therapy( ie during the first 96 hours)
  The development of persistently low blood pressure despite adequate measures to maintain normal blood pressure will be assessed and recorded throughout the hypothermia therapy.
Pulmonary Hemorrhage | Duration of hospital stay, an expected average of up to 4 weeks
  The development of Pulmonary hemorrhage at any stage during the patient's hospital stay will be recorded.
Intracranial Hemorrhage | Duration of hospital stay, an expected average of up to 4 weeks
  The development of Intracranial Hemorrhage at any stage during the patient's hospital stay will be recorded by serial head ultrasounds on day 1 , day 3 and as required.
Pulmonary Hypertension | Duration of Hypothermia therapy (ie during the first 96 hours)
  The development of pulmonary hypertension at any stage during the patient's hospital stay will be recorded.
Prolonged Blood Coagulation time | Duration of hypothermia therapy ( ie during the first 96 hours)
  The development of abnormal coagulation profile during hypothermia therapy will be recorded.
Culture Proven sepsis | Duration of hospital stay, an expected average of up to 4 weeks
  The development of sepsis with a positive blood culture during the patient's hospital stay will be recorded.
Necrotizing enterocolitis | Duration of hospital stay, an expected average of up to 4 weeks
  The development of necrotizing enterocolitis during the patient's hospital stay will be recorded.
Cardiac Arrhythmias | Duration of hypothermia therapy (ie during the first 96 hours)
  The development ofcardiac arrythmia during hypothermia therapy will be recorded.
Thrombocytopenia | Duration of hypothermia therapy (ie during the first 96 hours)
  The development of low platelet count (<20,000) during hypothermia therapy will be recorded
Major venous thrombosis | Duration of hospital stay, an expected average of up to 4 weeks
  The development of major venous thrombosis or a major vein thrombus during the patient's hospital stay will be recorded.
Renal Failure | Duration of hospital stay, an expected average of up to 4 weeks
  The development of renal failure during the patient's hospital stay will be recorded
Abnormal liver funcion tests (elevated liver enzymes) | Duration of hospital stay, an expected average of up to 4 weeks
  The devlopment of raised liver enzymes during the patient's hospital stay will be recorded.
Pneumonia | Duration of hospital stay, an expected average of up to 4 weeks
  The development of pneumonia during the patient's hospital stay will be assessed and recorded.
Pulmonary air leak syndrome | Duration of hospital stay, an expected average of up to 4 weeks
  The development of pulmonary air leak syndrome during the patient's hospital stay will be recorded.
Prolonged vs shortened hospital stay | First day of NICU admission till the day of discharge, an expected average of up to 4 weeks
  The entire duration of hopital stay will be assessed
Neurodevelopment score | On the day of discharge from hospital, an expected average of 4 weeks after admission
  A developmental paediatrician blinded to the study groups will assess the patient's neurodevlopment on the day of his or her discharge.
Abnormal aEEG | Before randomization and during hypothermia therapy (0 hours till 96 hours)
  The aEEG is used to measure the severity of Hypoxic Ischemic Encephalopathy (moderate or severe).
Presence of multiple handicaps | 18-24 months of age
  Multiple handicaps (( defined as the presence of any two of the following in an infant at the age of 18-24 months: neuromotor disability (level 3-5 on GMF Classification), mental delay (Bayley MDI score <70),epilepsy, cortical visual impairment, sensorineural hearing loss)).
Bayley Psychomotor Development Score less than 70 | 18-24 months of age
Sensorineural hearing loss equal to, or more than, 40 dB | 18-24 months of age
Epilepsy | 18-24 months of age
  Epilepsy is defined as recurrent seizures beyond the neonatal period, requiring anticonvulsant therapy at the time of assessment
Microcephaly | 18-24 months of age
  Defined as Head circumference more than 2 standard deviations below the mean
Result of EEG or MRI | within the first 14 days of life
  To moniter any abnormal EEG patterns and any evidence of Ischemic/Hemorrhagic lesions on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Sajjad Ur Rahman, MBBS.DCH.MCPS.FCPS.FRCPCH.FNP, Principal Investigator — Hamad Medical Corporation
Locations (7):
- Mansoura University Children's Hospital, Al Mansurah, Egypt
- University Malaya Medical Center (UMMC), Kuala Lumpur, Malaysia
- NICU,Women's Hospital, Hamad Medical Corporation, Doha, Baladīyat ad Dawḩah, Qatar
- Arrayan Hospital-Dr Sulaiman Al Habib Medical Group, Riyadh, Riyadh Region, Saudi Arabia
- Turkey (Türkiye) (2):
  - Zekai Tahir Burak Maternity Teaching Hospital, Ankara
  - Diyarbakir Children's Hospital, Diyarbakır
- Tawam Hospital, AlAin, United Arab Emirates

REFERENCES:
- [Background] Paul VK. Neonatal morbidity and mortality: report of the national neonatal and perinatal database. Indian Pediatr. 1999 Feb;36(2):167-9. No abstract available. PMID 10713810
- [Background] Bhat MA, Shah ZA, Makhdoomi MS, Mufti MH. Theophylline for renal function in term neonates with perinatal asphyxia: a randomized, placebo-controlled trial. J Pediatr. 2006 Aug;149(2):180-4. doi: 10.1016/j.jpeds.2006.03.053. PMID 16887430
- [Background] Paneth N. The causes of cerebral palsy. Recent evidence. Clin Invest Med. 1993 Apr;16(2):95-102. PMID 8513618
- [Background] Dixon G, Badawi N, Kurinczuk JJ, Keogh JM, Silburn SR, Zubrick SR, Stanley FJ. Early developmental outcomes after newborn encephalopathy. Pediatrics. 2002 Jan;109(1):26-33. doi: 10.1542/peds.109.1.26. PMID 11773538
- [Background] Edwards AD, Azzopardi DV. Hypothermic neural rescue: work continues. J Pediatr. 2010 Sep;157(3):351-2. doi: 10.1016/j.jpeds.2010.06.029. Epub 2010 Jul 24. No abstract available. PMID 20659738
- [Background] Gluckman PD, Wyatt JS, Azzopardi D, Ballard R, Edwards AD, Ferriero DM, Polin RA, Robertson CM, Thoresen M, Whitelaw A, Gunn AJ. Selective head cooling with mild systemic hypothermia after neonatal encephalopathy: multicentre randomised trial. Lancet. 2005 Feb 19-25;365(9460):663-70. doi: 10.1016/S0140-6736(05)17946-X. PMID 15721471
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Background] Simbruner G, Mittal RA, Rohlmann F, Muche R; neo.nEURO.network Trial Participants. Systemic hypothermia after neonatal encephalopathy: outcomes of neo.nEURO.network RCT. Pediatrics. 2010 Oct;126(4):e771-8. doi: 10.1542/peds.2009-2441. Epub 2010 Sep 20. PMID 20855387
- [Background] Zhou WH, Cheng GQ, Shao XM, Liu XZ, Shan RB, Zhuang DY, Zhou CL, Du LZ, Cao Y, Yang Q, Wang LS; China Study Group. Selective head cooling with mild systemic hypothermia after neonatal hypoxic-ischemic encephalopathy: a multicenter randomized controlled trial in China. J Pediatr. 2010 Sep;157(3):367-72, 372.e1-3. doi: 10.1016/j.jpeds.2010.03.030. Epub 2010 May 20. PMID 20488453
- [Background] Levene MI. Cool treatment for birth asphyxia, but what's next? Arch Dis Child Fetal Neonatal Ed. 2010 May;95(3):F154-7. doi: 10.1136/adc.2009.165738. No abstract available. PMID 20444808
- [Background] Jacobs S, Hunt R, Tarnow-Mordi W, Inder T, Davis P. Cooling for newborns with hypoxic ischaemic encephalopathy. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003311. doi: 10.1002/14651858.CD003311.pub2. PMID 17943788
- [Background] Edwards AD, Brocklehurst P, Gunn AJ, Halliday H, Juszczak E, Levene M, Strohm B, Thoresen M, Whitelaw A, Azzopardi D. Neurological outcomes at 18 months of age after moderate hypothermia for perinatal hypoxic ischaemic encephalopathy: synthesis and meta-analysis of trial data. BMJ. 2010 Feb 9;340:c363. doi: 10.1136/bmj.c363. PMID 20144981
- [Background] Rutherford M, Ramenghi LA, Edwards AD, Brocklehurst P, Halliday H, Levene M, Strohm B, Thoresen M, Whitelaw A, Azzopardi D. Assessment of brain tissue injury after moderate hypothermia in neonates with hypoxic-ischaemic encephalopathy: a nested substudy of a randomised controlled trial. Lancet Neurol. 2010 Jan;9(1):39-45. doi: 10.1016/S1474-4422(09)70295-9. Epub 2009 Nov 5. PMID 19896902
- [Background] Rouse DJ, Hirtz DG, Thom E, Varner MW, Spong CY, Mercer BM, Iams JD, Wapner RJ, Sorokin Y, Alexander JM, Harper M, Thorp JM Jr, Ramin SM, Malone FD, Carpenter M, Miodovnik M, Moawad A, O'Sullivan MJ, Peaceman AM, Hankins GD, Langer O, Caritis SN, Roberts JM; Eunice Kennedy Shriver NICHD Maternal-Fetal Medicine Units Network. A randomized, controlled trial of magnesium sulfate for the prevention of cerebral palsy. N Engl J Med. 2008 Aug 28;359(9):895-905. doi: 10.1056/NEJMoa0801187. PMID 18753646
- [Background] Bhat MA, Charoo BA, Bhat JI, Ahmad SM, Ali SW, Mufti MU. Magnesium sulfate in severe perinatal asphyxia: a randomized, placebo-controlled trial. Pediatrics. 2009 May;123(5):e764-9. doi: 10.1542/peds.2007-3642. Epub 2009 Apr 6. PMID 19349375